CLINICAL TRIAL: NCT04604353
Title: Early Detection of Coronary Artery Disease by Polygenic and Metabolic Risk Scoring in at Risk Patients: Comparison With Coronary Computed Tomography
Brief Title: Early Detection of Coronary Artery Disease by Polygenic and Metabolic Risk Scoring
Acronym: EDCAD-PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 492/20
Record Dates: First submitted 2020-10-19; First posted 2020-10-27 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Randomization to provision of PRS-based or CCS-based risk
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will receive baseline and 12 month risk based on Pooled Cohort Equation and photographic evidence of treatment adherence
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRS score group (Experimental): Risk information provided on the basis of Polygenic Risk Score combined with the Pooled Cohort Equation
  Interventions: Diagnostic Test: Polygenic Risk Score
- CCS score group (Active Comparator): Risk information provided on the basis of Coronary Calcium Score combined with the Pooled Cohort Equation
  Interventions: Diagnostic Test: Coronary Calcium Score

INTERVENTIONS:
Diagnostic Test: Polygenic Risk Score — Risk description to patient based on PRS
  Arms: PRS score group
Diagnostic Test: Coronary Calcium Score — Risk description to patient based on CCS
  Arms: CCS score group

SUMMARY:
The overall goal of this study is to develop a combined polygenic risk score (PRS) and metabolic risk score (MRS) and determine its impact on selecting community members for CCS. The trial component of this study will compare the use of these scores to motivate people to adhere to therapy, an ongoing challenge for clinicians, by providing feedback in a meaningful form to both the clinicians and the patients.

DETAILED DESCRIPTION:
Patients undergoing a polygenic risk score (PRS), metabolic risk score (MRS) and coronary calcium score (CCS) will be randomized to receive PRS and CCS information and followed for the reduction of risk over 12 months. This information will provide information about how to motivate people to adhere to therapy, by providing feedback in a meaningful form to both the clinicians and the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Asymptomatic subjects age 40-70y
2. Statin naïve
3. TC ≤ 6.5 mmol/L and LDLC <5 mmol/L, and
4. 5 year Australian risk ≥2%.

Exclusion Criteria:

1. Symptomatic coronary, cerebrovascular, or peripheral vascular disease
2. Intolerance of statins or currently on statins for any length of time
3. Pre-existing muscle disease (eg polymyositis, fibromyalgia) - this may be confused with myalgia from statins
4. Patients on drugs that increase the risk of myopathy/rhabdomyolysis such as cyclosporine and strong CYP3A4 inhibitors (e.g., clarithromycin, itraconazole, and HIV/hepatitis C protease inhibitors)
5. Atrial fibrillation (interferes with CTCA)
6. Chronic kidney disease on haemodialysis (because of vascular calcification) or GFR <50ml/min per 1.73m2 using the Modification of Diet in Renal Disease (MDRD) formula
7. Inability to provide informed consent
8. Major systemic illness eg. malignancy; rheumatoid arthritis
9. Women of child bearing potential (due to performance of CT)
10. Poorly controlled hypertension: SBP> 200 and or DBP > 100
11. Severe psychiatric disorder (eg bipolar depression; psychosis)
12. Patients eligible for treatment based on current Australian guidelines (5 year risk >15%)
13. Patients eligible for treatment based on current PBS thresholds TC >7.5 mmol/l and other criteria (see below).

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2020-12-07 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in cardiovascular risk in each group | 12 months
  Change in cardiovascular risk (expressed as pooled cohort equation 10-year risk percentage) from baseline to follow-up

SECONDARY OUTCOMES:
Medication adherence in each group | 12 months
  Proportion of lipid-lowering tablets taken

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Marwick, MD, PhD, MPH, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Data sharing based available on application to the study PI